CLINICAL TRIAL: NCT02613403
Title: A Phase II, Randomized, Open-Label Clinical Trial to Study the Efficacy and Safety of the Combination Regimen of MK-3682B (MK-5172 + MK-3682 + MK-8408 Fixed Dose Combination (FDC)) in Subjects With Chronic HCV GT1 or GT3 Infection Who Have Failed a Direct Acting Antiviral Regimen
Brief Title: Efficacy and Safety of Grazoprevir (+) Uprifosbuvir (+) Ruzasvir (MK-3682B) (MK-5172 + MK-3682 + MK-8408) Fixed Dose Combination in Chronic HCV Participants Failing Prior Antiviral Treatment (MK-3682-021)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3682-021; MK-3682-021 (Other: Merck Protocol Number); 2015-001483-19 (EudraCT Number)
Record Dates: First submitted 2015-11-20; First posted 2015-11-24 (Estimated); Results first posted 2018-03-20 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Hepatitis; Hepatitis C; Digestive System Diseases; Flaviviridae Infections; Hepatitis, Viral, Human; Liver Diseases; RNA Virus Infections; Virus Diseases
MeSH Terms: conditions — Hepatitis; Hepatitis C; Digestive System Diseases; Flaviviridae Infections; Hepatitis, Viral, Human; Liver Diseases; RNA Virus Infections; Virus Diseases | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- [Part A, Arm 1] Prior SOF/LDV Failure: MK-3682B + RBV (Experimental): C or NC HCV GT1 participants previously failing a DAA regimen of SOF/LDV receive MK-3682B, an FDC of GZR (MK-5172 [50 mg]) + UPR (MK-3682 [225 mg]) + RZR (MK-8408 [30 mg]), administered as 2 tablets once daily in combination with RBV twice daily for 16 weeks.
  Interventions: Drug: MK-3682B; Drug: Ribavirin
- [Part A, Arm 2] Prior SOF/LDV Failure: MK-3682B (Experimental): C or NC HCV GT1 participants previously failing a DAA regimen of SOF/LDV receive MK-3682B, an FDC of GZR (MK-5172 [50 mg]) + UPR (MK-3682 [225 mg]) + RZR (MK-8408 [30 mg]), administered as 2 tablets once daily for 24 weeks.
  Interventions: Drug: MK-3682B
- [Part A, Arm 3] Prior GZR/EBR Failure: MK-3682B + RBV (Experimental): C or NC HCV GT1 participants previously failing a DAA regimen of GZR/EBR (MK-5172/MK-8742) receive MK-3682B, an FDC of GZR (MK-5172 [50 mg]) + UPR (MK-3682 [225 mg]) + RZR (MK-8408 [30 mg]), administered as 2 tablets once daily in combination with RBV twice daily for 16 weeks.
  Interventions: Drug: MK-3682B; Drug: Ribavirin
- [Part A, Arm 4] Prior GZR/EBR Failure: MK-3682B (Experimental): C or NC HCV GT1 participants previously failing a DAA regimen of GZR/EBR (MK-5172/MK-8742) receive MK-3682B, an FDC of GZR (MK-5172 [50 mg]) + UPR (MK-3682 [225 mg]) + RZR (MK-8408 [30 mg]), administered as 2 tablets once daily for 24 weeks.
  Interventions: Drug: MK-3682B
- [Part B] Prior DAA (GT1-6) or SOF/PR (GT3) Failure: MK-3682B (Experimental): C or NC HCV participants previously failing any all-oral DAA regimen (GT1-6) or SOF/PR regimen (GT 3 only) receive MK-3682B, an FDC of GZR (MK-5172 [50 mg]) + UPR (MK-3682 [225 mg]) + RZR (MK-8408 [30 mg]), administered as 2 tablets once daily for 16 weeks.
  Interventions: Drug: MK-3682B

INTERVENTIONS:
Drug: MK-3682B — Two MK- 3682B 1,136 mg FDC tablets each containing 50 mg MK-5172 (GZR), 225 mg MK-3682 (UPR, formerly IDX21437), and 30 mg MK-8408 (RZR) taken once daily by mouth.
Drug: Ribavirin — Ribavirin 200 mg capsules, taken twice daily by mouth as part of a weight-based dosing regimen. Depending on participant body weight, total daily dose of Ribavirin may be 800, 1000, 1200 or 1400 mg per day.
  Arms: [Part A, Arm 1] Prior SOF/LDV Failure: MK-3682B + RBV; [Part A, Arm 3] Prior GZR/EBR Failure: MK-3682B + RBV

SUMMARY:
This is a randomized, multicenter, 2-part, open-label trial of the combination regimen of grazoprevir (GZR [MK-5172]; 100mg), uprifosbuvir (UPR [MK-3682]; 450 mg) and ruzasvir (RZR [MK-8408]; 60 mg) with and without Ribavirin (RBV) in cirrhotic (C) or non-cirrhotic (NC) participants infected with hepatitis C virus (HCV) previously failing a direct-acting antiviral regimen (DAA). The combination regimen, referred to as MK-3682B, will be administered as two fixed-dose combination (FDC) tablets, given once-daily. The study will evaluate the efficacy of MK-3682B with or without RBV as assessed by the proportion of participants achieving Sustained Virologic Response 12 weeks (SVR12) after the end of all study therapy.

DETAILED DESCRIPTION:
This trial was divided into Part A and Part B. In Part A, comprised of 4 treatment arms, C or NC participants with HCV genotype (GT) 1 infection previously failing a DAA regimen of either sofosbuvir (SOF)/ledipasvir (LDV) [Arms 1 and 2] or elbasvir (EBR)/GZR [Arms 3 and 4] were randomized to receive either one of the following: 1) MK-3682B + RBV for 16 weeks [Arms 1 and 3]; or 2) MK-3682B for 24 weeks [Arms 2 and 4]. Study Part A was completed as planned per study protocol. In Part B, C or NC participants with GT1 through GT6 infection previously failing any all-oral DAA regimen (GT1-6) or SOF/pegylated interferon and ribavirin (PR) regimen (GT 3 only) were to receive MK-3682B for 16 weeks. However, the trial was terminated prior to participant enrollment for study Part B.

Participants in MK-5172-017 (NCT01667081) were eligible for enrollment in the study.

ELIGIBILITY:
Inclusion Criteria:

Part A

* Has documented chronic HCV GT1 or HCV GT3 infection with no evidence of non-typeable or mixed genotype.
* Has documented relapse, defined as having HCV RNA target not detected at end-of-treatment, but HCV RNA quantifiable during follow-up, after treatment with one of the following DAA regimens either by approved dosage and duration or by completion of a clinical trial: GT1: SOF/LDV ± RBV; GT1: GZR/EBR ± RBV; GT3: SOF + RBV; GT3: SOF + PR; GT3: SOF + DCV ± RBV; GT3: SOF/LDV ± RBV.
* Is otherwise healthy.
* If male, be not of reproductive potential or agree to avoid impregnating a partner beginning at least 2 weeks prior to administration of the initial dose of study drug, through 6 months after taking the last dose of study drug (or longer if dictated by local regulations), by complying with one of the following: (1) practice abstinence from heterosexual activity or (2) use (or have their partner use) two forms of acceptable contraception during heterosexual activity which may include oral contraceptives.

Part B

* Has documented chronic HCV GT1, GT2, GT3, GT4, GT5, GT6 infection with no evidence of non-typeable or mixed genotype.
* Has documented virologic failure, defined as having quantifiable HCV RNA at any time after completion of HCV therapy with a DAA regimen either by approved dosage and duration or by completion of a clinical trial that was not attributed to re-infection: GT1, GT2, GT4, GT5, or GT6: any prior all-oral DAA regimens; GT3: any prior all-oral DAA regimen or SOF/PR. Participants [Parts A and B] who previously failed PR treatment, with or without simepravir (SIM), boceprevir (BOC), or telaprevir (TPV), prior to receiving DAA therapy, may also be enrolled.

Parts A and B

* Has HCV RNA ≥ 10,000 IU/mL in peripheral blood at enrollment.
* Has either absence of cirrhosis or presence of compensated cirrhosis.
* If female, be not of reproductive potential or agree to avoid becoming pregnant beginning at least 2 weeks prior to administration of the initial dose of study drug, through either 6 months [Part A] or 14 days [Part B] after taking the last dose of study drug (or longer if dictated by local regulations), by complying with one of the following: (1) practice abstinence from heterosexual activity or (2) use (or have their partner use) two forms of acceptable contraception during heterosexual activity which may include oral contraceptives.
* For HIV co-infected participants: 1) have documented HIV-1 infection [Part A] or HIV infection [Part B]; 2) either not be currently on antiretroviral therapy (ART) with no plans to initiate ART while participating in this study or have well controlled HIV on ART; and 3) have at least one viable antiretroviral regimen alternative beyond their current regimen in the event of HIV virologic failure and the development of anti-retroviral drug resistance [Part A].

Exclusion Criteria:

Part A

* Has previously received a DAA containing regimen other than the permitted regimens listed above.
* Did not complete their prior DAA therapy due to intolerance to the DAA regimen or who failed the DAA regimen for reasons other than relapse (e.g., virologic breakthrough, rebound or non-response, non-compliance, lost to follow-up, withdrew consent).
* Is a male whose female partner(s) is/are pregnant or is a male who is expecting to donate sperm or planning to impregnate female partner(s) from at least two weeks prior to Day 1 through at least 6 months after last dose of study drug, or longer if dictated by local regulations.
* Has personal or family history of Torsade de pointes.
* Has chronic pulmonary disease.
* Has an hemoglobinopathy.
* Has central nervous system (CNS) trauma requiring intubation, intracranial pressure monitoring, brain meningeal or skull surgery, or resulting in seizure, coma, permanent neurologic deficits, abnormal brain imaging, or cerebral spinal fluid (CSF) leak; prior brain hemorrhage and/or intracranial aneurysms (whether adequately repaired or not).
* Has current or history of seizure disorder unless seizure was >10 years ago, a single isolated event, no history of or current use of anti-seizure medications, and a documented normal neurological examination at Day 1.
* Has history of stroke or transient ischemic attack.

Part B

* Did not complete their prior DAA therapy due to intolerance to the DAA regimen or who failed the DAA regimen for reasons other than virologic failure.
* Has any major medical condition, clinically-significant illness (other than HCV), pretrial laboratory or ECG abnormality, or history of any illness that might interfere with treatment, assessment, compliance or pose additional risk in administering study drug to the participant.

Parts A and B

* Is under the age of legal consent, is mentally or legally incapacitated, has significant emotional problems at the time of pre-study screening visit or expected during the conduct of the study or has a history of a clinically significant psychiatric disorder which, in the opinion of the investigator, would interfere with the study procedures.
* Has evidence of decompensated liver disease manifested by the presence of or history of ascites, esophageal or gastric variceal bleeding, hepatic encephalopathy or other signs or symptoms of advanced liver disease.
* Has cirrhosis classified as Child-Pugh Class B or C or has a Pugh-Turcotte score >6
* Is co-infected with hepatitis B virus (HBV)
* For participants with HIV, has a history of opportunistic infection in the 6 months prior to screening.
* Has a history of malignancy ≤5 years prior to enrollment except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer or carcinoma in situ; or is under evaluation for other active or suspected malignancy.
* Has cirrhosis and liver imaging within 6 months of Day 1 showing evidence of hepatocellular carcinoma (HCC) or is under evaluation for HCC.
* Is currently participating or has participated in a study with an investigational compound within 30 days of signing informed consent and is not willing to refrain from participating in another such study during the course of this study (trial treatment period). Participants participating in MK-5172-017 (NCT01667081) may be enrolled in this study, MK- 3682-021.
* Has clinically-relevant drug or alcohol abuse within 12 months of screening
* Is a female and is pregnant or breastfeeding or expecting to conceive or donate eggs from at least 2 weeks prior to Day 1 through at least 6 months [Part A] or 14 days [Part B] after last dose of study drug, or longer if dictated by local regulations.
* Has organ transplants (including hematopoietic stem cell transplants) other than cornea and hair.
* Has history of gastric surgery or history of malabsorption disorders.
* Has current or history of any clinically significant cardiac abnormalities/dysfunction.
* Has medical/surgical conditions that may result in a need for hospitalization during the period of the study.
* Has a medical condition requiring, or likely to require, chronic systemic administration of corticosteroids, tumor necrosis factor (TNF) antagonists, or other immunosuppressant drugs during the course of the study
* Has evidence of history of chronic hepatitis not caused by HCV. Participants with history of acute non-HCV-related hepatitis, that resolved >6 months before study entry, may be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2015-12-10 (Actual); Primary Completion 2017-01-09 (Actual); Study Completion 2017-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Wyles D, Wedemeyer H, Ben-Ari Z, Gane EJ, Hansen JB, Jacobson IM, Laursen AL, Luetkemeyer A, Nahass R, Pianko S, Zeuzem S, Jumes P, Huang HC, Butterton J, Robertson M, Wahl J, Barr E, Joeng HK, Martin E, Serfaty L; C-CREST Part C and C-SURGE Investigators. Grazoprevir, ruzasvir, and uprifosbuvir for hepatitis C virus after NS5A treatment failure. Hepatology. 2017 Dec;66(6):1794-1804. doi: 10.1002/hep.29358. Epub 2017 Oct 30. PMID 28688129

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For study Part A, 94 cirrhotic (C) or non-cirrhotic (NC) participants with chronic hepatitis C virus (HCV) genotype (GT) 1 previously failing a direct-acting antiviral regimen (DAA) were randomized, with 1 participant withdrawing prior to receiving study treatment.
  The trial was terminated prior to participant enrollment for study Part B.
Groups:
- [Part A, Arm 1] Prior SOF/LDV Failure: MK-3682B + RBV: C or NC HCV GT1 participants previously failing a DAA regimen of sofosbuvir (SOF)/ledipasvir (LDV) receive MK-3682B, a fixed dose combination (FDC) of grazoprevir (GZR; MK-5172 [50 mg]) + uprifosbuvir (UPR; MK-3682 [225 mg]) + ruzasvir (RZR; MK-8408 [30 mg]), administered as 2 tablets once daily in combination with ribavirin (RBV) twice daily for 16 weeks.
- [Part A, Arm 3] Prior GZR/EBR Failure: MK-3682B + RBV: C or NC HCV GT1 participants previously failing a DAA regimen of GZR/elbasvir (EBR) (MK-5172/MK-8742) receive MK-3682B, an FDC of GZR (MK-5172 [50 mg]) + UPR (MK-3682 [225 mg]) + RZR (MK-8408 [30 mg]), administered as 2 tablets once daily in combination with RBV twice daily for 16 weeks.
- [Part B] Prior DAA (GT1-6) or SOF/PR (GT3) Failure: MK-3682B: C or NC HCV participants previously failing any all-oral DAA regimen (GT1-6) or SOF/pegylated interferon and ribavirin (PR) regimen (GT 3 only) receive MK-3682B, an FDC of GZR (MK-5172 [50 mg]) + UPR (MK-3682 [225 mg]) + RZR (MK-8408 [30 mg]), administered as 2 tablets once daily for 16 weeks.
Period: Overall Study
Arm/Group | [Part A, Arm 1] Prior SOF/LDV Failure: MK-3682B + RBV | [Part A, Arm 2] Prior SOF/LDV Failure: MK-3682B | [Part A, Arm 3] Prior GZR/EBR Failure: MK-3682B + RBV | [Part A, Arm 4] Prior GZR/EBR Failure: MK-3682B | [Part B] Prior DAA (GT1-6) or SOF/PR (GT3) Failure: MK-3682B
Started | 36 | 36 | 9 | 13 | 0 (Study terminated prior to participant recruitment for study Part B.)
Treated | 35 | 36 | 9 | 13 | 0 (Study terminated prior to participant recruitment for study Part B.)
Completed | 34 | 35 | 9 | 13 | 0 (Study terminated prior to participant recruitment for study Part B.)
Not Completed | 2 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Includes only randomized participants in Study Part A receiving ≥1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | [Part A, Arm 1] Prior SOF/LDV Failure: MK-3682B + RBV | [Part A, Arm 2] Prior SOF/LDV Failure: MK-3682B | [Part A, Arm 3] Prior GZR/EBR Failure: MK-3682B + RBV | [Part A, Arm 4] Prior GZR/EBR Failure: MK-3682B | Total
Number analyzed (Participants) | 35 | 36 | 9 | 13 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (8.4) | 58.9 (6.6) | 57.3 (8.5) | 53.9 (11.0) | 58.1 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 3 | 4 | 13
  Male | 31 | 34 | 6 | 9 | 80

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virologic Response 12 Weeks After The End of Study Therapy (SVR12)
Description: The percentage of participants achieving SVR12 was determined, defined as having a plasma HCV ribonucleic acid (RNA) level below the lower limit of quantification (LLOQ) 12 weeks after the end of study therapy. Plasma HCV RNA level was measured using the Roche COBAS™ AmpliPrep/COBAS™ Taqman™ HCV Test, v2.0 ® assay with a LLOQ of 15 IU/mL.
Time Frame: 12 weeks following final dose of study treatment ([MK-3682B + RBV Groups]: Study Week 28; [MK-3682B Groups]: Study Week 36)
Population: All randomized participants in Part A receiving ≥1 dose of study treatment. Part B was terminated prior to participant enrollment and was not included for analysis.
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | [Part A, Arm 1] Prior SOF/LDV Failure: MK-3682B + RBV | [Part A, Arm 2] Prior SOF/LDV Failure: MK-3682B | [Part A, Arm 3] Prior GZR/EBR Failure: MK-3682B + RBV | [Part A, Arm 4] Prior GZR/EBR Failure: MK-3682B
Number analyzed (Participants) | 35 | 36 | 9 | 13
Percentage | 97.1 [85.1 to 99.9] | 100.0 [90.3 to 100.0] | 100.0 [66.4 to 100.0] | 100.0 [75.3 to 100.0]

2. Primary Outcome: Number of Participants Who Experienced an Adverse Event
Description: The number of participants experiencing an adverse event (AE) was assessed. An AE is any unfavorable and unintended medical occurrence, symptom, or disease witnessed in a participant, regardless of whether or not a causal relationship with the study treatment can be demonstrated. Further, any worsening of a preexisting condition that is temporally associated with the use of the study treatment is also considered an AE.
Time Frame: Up to 2 weeks following cessation of study treatment ([MK-3682B + RBV Groups]: Up to Week 18; [MK-3682B Groups]: Up to Week 26)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | [Part A, Arm 1] Prior SOF/LDV Failure: MK-3682B + RBV | [Part A, Arm 2] Prior SOF/LDV Failure: MK-3682B | [Part A, Arm 3] Prior GZR/EBR Failure: MK-3682B + RBV | [Part A, Arm 4] Prior GZR/EBR Failure: MK-3682B
Number analyzed (Participants) | 35 | 36 | 9 | 13
Participants | 31 | 27 | 9 | 12

3. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an Adverse Event
Description: The number of participants discontinuing study drug due to an AE was assessed.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | [Part A, Arm 1] Prior SOF/LDV Failure: MK-3682B + RBV | [Part A, Arm 2] Prior SOF/LDV Failure: MK-3682B | [Part A, Arm 3] Prior GZR/EBR Failure: MK-3682B + RBV | [Part A, Arm 4] Prior GZR/EBR Failure: MK-3682B
Number analyzed (Participants) | 35 | 36 | 9 | 13
Participants | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants Who Experienced a Serious Adverse Event
Description: The number of participants experiencing a serious adverse event (SAE) was assessed. An SAE is an adverse event that: results in death; is life threatening; results in persistent or significant disability or incapacity; results in or prolongs a hospitalization; is a congenital anomaly or birth defect; is a cancer; or may jeopardize the participant, potentially require medical or surgical intervention.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | [Part A, Arm 1] Prior SOF/LDV Failure: MK-3682B + RBV | [Part A, Arm 2] Prior SOF/LDV Failure: MK-3682B | [Part A, Arm 3] Prior GZR/EBR Failure: MK-3682B + RBV | [Part A, Arm 4] Prior GZR/EBR Failure: MK-3682B
Number analyzed (Participants) | 35 | 36 | 9 | 13
Participants | 3 | 4 | 0 | 1

5. Primary Outcome: Number of Participants Who Experienced a Drug-Related Adverse Event
Description: The number of participants experiencing a drug-related AE was assessed. A drug-related AE was an AE thought to be possibly, probably, or definitely related to the study drug as determined by the investigator.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | [Part A, Arm 1] Prior SOF/LDV Failure: MK-3682B + RBV | [Part A, Arm 2] Prior SOF/LDV Failure: MK-3682B | [Part A, Arm 3] Prior GZR/EBR Failure: MK-3682B + RBV | [Part A, Arm 4] Prior GZR/EBR Failure: MK-3682B
Number analyzed (Participants) | 35 | 36 | 9 | 13
Participants | 23 | 18 | 9 | 5

6. Primary Outcome: Number of Participants Who Experienced a Serious and Drug-Related Adverse Event
Description: The number of participants experiencing a serious and drug-related AE was assessed.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | [Part A, Arm 1] Prior SOF/LDV Failure: MK-3682B + RBV | [Part A, Arm 2] Prior SOF/LDV Failure: MK-3682B | [Part A, Arm 3] Prior GZR/EBR Failure: MK-3682B + RBV | [Part A, Arm 4] Prior GZR/EBR Failure: MK-3682B
Number analyzed (Participants) | 35 | 36 | 9 | 13
Participants | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants Who Experienced an Accidental or Intentional Overdose Without Adverse Effect
Description: The number of participants experiencing an accidental or intentional overdose without adverse effect was determined. Per study protocol, any occurrence of a participant receiving either MK-3682B or RBV at any dose higher than prescribed was considered an overdose. If this definition of overdose was met without any associated clinical symptoms or abnormal laboratory results, this occurrence of overdose was reported as an accidental or intentional overdose without adverse effect.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | [Part A, Arm 1] Prior SOF/LDV Failure: MK-3682B + RBV | [Part A, Arm 2] Prior SOF/LDV Failure: MK-3682B | [Part A, Arm 3] Prior GZR/EBR Failure: MK-3682B + RBV | [Part A, Arm 4] Prior GZR/EBR Failure: MK-3682B
Number analyzed (Participants) | 35 | 36 | 9 | 13
Participants | 1 | 3 | 2 | 1

8. Primary Outcome: Number of Participants Who Experienced a Non-Overdose Event of Clinical Interest
Description: The number of participants experiencing a non-overdose event of clinical interest (ECI) was determined. Non-overdose ECIs, assessed from initiation of study therapy through 14 days following study treatment cessation, included the following: 1) aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >500 IU/L; or 2) AST or ALT >3x nadir value and >3X upper limit normal (ULN).
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | [Part A, Arm 1] Prior SOF/LDV Failure: MK-3682B + RBV | [Part A, Arm 2] Prior SOF/LDV Failure: MK-3682B | [Part A, Arm 3] Prior GZR/EBR Failure: MK-3682B + RBV | [Part A, Arm 4] Prior GZR/EBR Failure: MK-3682B
Number analyzed (Participants) | 35 | 36 | 9 | 13
Participants | 0 | 1 | 0 | 0

9. Primary Outcome: Number of Participants Who Experienced AST/ALT >5x Upper Limit Normal (ULN)
Description: The number of participants experiencing AST / ALT >5 times ULN from study week 4 until 2 weeks following completion of study therapy was determined.
Time Frame: From Study Week 4 up to 2 weeks following cessation of study treatment ([MK-3682B + RBV Groups]: Up to Week 18; [MK-3682B Groups]: Up to Week 26)
Population: All randomized participants in Part A receiving ≥1 dose of study treatment with ≥1 AST/ALT measurement subsequent to study week 4. One participant with prior SOF/LDV failure receiving MK-3682B + RBV withdrew from study before study week 4 and was excluded from analysis. Part B terminated prior to enrollment and was not included for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | [Part A, Arm 1] Prior SOF/LDV Failure: MK-3682B + RBV | [Part A, Arm 2] Prior SOF/LDV Failure: MK-3682B | [Part A, Arm 3] Prior GZR/EBR Failure: MK-3682B + RBV | [Part A, Arm 4] Prior GZR/EBR Failure: MK-3682B
Number analyzed (Participants) | 34 | 36 | 9 | 13
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 2 weeks following cessation of study treatment ([MK-3682B + RBV Groups]: Up to Week 18; [MK-3682B Groups]: Up to Week 26)
Description: Includes only randomized participants in Study Part A receiving ≥1 dose of study treatment. The trial was terminated prior to participant enrollment for study Part B.
Arm/Group | [Part A, Arm 1] Prior SOF/LDV Failure: MK-3682B + RBV | [Part A, Arm 2] Prior SOF/LDV Failure: MK-3682B | [Part A, Arm 3] Prior GZR/EBR Failure: MK-3682B + RBV | [Part A, Arm 4] Prior GZR/EBR Failure: MK-3682B
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/36 | 0/9 | 0/13
Serious Adverse Events (participants affected / at risk) | 3/35 | 4/36 | 0/9 | 1/13
Other Adverse Events (participants affected / at risk) | 29/35 | 25/36 | 9/9 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | [Part A, Arm 1] Prior SOF/LDV Failure: MK-3682B + RBV (N=35) | [Part A, Arm 2] Prior SOF/LDV Failure: MK-3682B (N=36) | [Part A, Arm 3] Prior GZR/EBR Failure: MK-3682B + RBV (N=9) | [Part A, Arm 4] Prior GZR/EBR Failure: MK-3682B (N=13)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | [Part A, Arm 1] Prior SOF/LDV Failure: MK-3682B + RBV (N=35) | [Part A, Arm 2] Prior SOF/LDV Failure: MK-3682B (N=36) | [Part A, Arm 3] Prior GZR/EBR Failure: MK-3682B + RBV (N=9) | [Part A, Arm 4] Prior GZR/EBR Failure: MK-3682B (N=13)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 3 (4) | 2 (2) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 15 (17) | 7 (7) | 6 (10) | 5 (5)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 3 (4) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (3) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 2 (2) | 1 (1)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 5 (5) | 5 (7) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Emotional disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (4) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (6) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 6 (8) | 2 (2) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.